CLINICAL TRIAL: NCT06173466
Title: Thoracic Paravertebral Block With Liposomal Bupivacaine Versus Standard Bupivacaine Combined With Dexamethasone for Postoperative Analgesia in Patients Undergoing Liver Resection
Brief Title: Postoperative Analgesia With Liposomal Bupivacaine Versus Standard Bupivacaine Combined With Dexamethasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2023-941 (IIT)
Record Dates: First submitted 2023-11-30; First posted 2023-12-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Liver Cancer
Keywords: Liver Resection; Thoracic Paravertebral Block; Liposomal Bupivacaine
MeSH Terms: conditions — Liver Neoplasms | interventions — Dexamethasone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient were performed TPVB in preoperative room before surgery. And the patient, care provider, anesthesiologist in OR, investigator and outcome assessor were blind to the study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal bupivacaine (Experimental): Patients in the bupivacaine liposomal group were treated with liposome bupivacaine 133 mg under ultrasound-guided TPVB. And ultrasound-guided TPVB was performed at the right T7-8, T8-9, T9-10, and T10-11 paravertebral interval under left lateral decubitus position, with 7.5 ml of medication injected into each paravertebral interval, for a total of 30 ml.
  Interventions: Drug: Liposomal bupivacaine
- Standard bupivacaine combined with dexamethasone (Active Comparator): Patients in the standard control group were treated with 0.5% bupivacaine hydrochloride 150 mg combined with dexamethasone 4 mg. the volume were expended to 30ml in both groups with normal saline. And ultrasound-guided TPVB was performed at the right T7-8, T8-9, T9-10, and T10-11 paravertebral interval under left lateral decubitus position, with 7.5 ml of medication injected into each paravertebral interval, for a total of 30 ml.
  Interventions: Drug: Bupivacaine Hydrochloride combined with dexamethasone

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine 133mg was injected to paravertebral intervals of right T7/8, T8/9, T9//10, T10/11 via ultrasound-guided TPVB
  Other Names: LB group (experimental group)
  Arms: Liposomal bupivacaine
Drug: Bupivacaine Hydrochloride combined with dexamethasone — Standard bupivacaine combined with dexamethasone 4mg was injected to paravertebral intervals of right T7/8, T8/9, T9//10, T10/11 via ultrasound-guided TPVB
  Other Names: SB Group (control group)
  Arms: Standard bupivacaine combined with dexamethasone

SUMMARY:
Liposomal bupivacaine is a novel long-acting local anesthetic approved by the FDA for postoperative analgesia because of its ability to significantly prolong the analgesic effect for up to 72 hours. Up to now, no study has demonstrated the effect of postoperative analgesia with liposomal bupivacaine by thoracic paravertebral block (TPVB). The aim of this study was to evaluate the efficacy of liposomal bupivacaine for pain management and recovery after liver resection.

Methods: 96 patients were involved in this randomized, prospective, single-blind study. Patients with hepatocellular carcinoma who were undergoing liver resection were divided into two groups: liposome bupivacaine group (liposomal bupivacaine 133mg) and standard bupivacaine combined with dexamethasone group (standard bupivacaine 150mg and dexamethasone 5mg). Both groups were applied ultrasound guided TPVB. The primary outcome was the cumulative opioid consumptionfor 72 hours. Secodary outcomes included QoR-40 at 72 hours, pain visual analog scale (VAS) score area under the curve (AUC) from 6 hours to 3 months, sleep quality at 1 month and 3 months postoperatively. Adverse events and serious adverse events 3 months after TPVB were also recorded.

DETAILED DESCRIPTION:
After approved by the Ethics Committee of Zhejiang Cancer Hospital (approval number IRB-2023-941 (IIT)). The study was registered before patient enrollment in Clinicaltrials. Written informed consent was obtained from all participants. The study was performed anticipated from November 9, 2023 to Dec 31, 2025. 96 adult hepatocellular carcinoma patients aged 18-75 years, ASA physical state I and III, who underwent elective or limited partial hepatectomy without allergy to the study drugs were enrolled in this study.

Basic monitoring such as 3-lead electrocardiogram, pulse oximetry, and noninvasive blood pressure were arranged preoperatively. Patients in the bupivacaine liposome group were treated with liposome bupivacaine 133 mg, and patients in the standard control group were treated with 0.5% bupivacaine hydrochloride 150 mg combined with dexamethasone 4 mg, the volume were expended to 30ml in both groups with normal saline. And ultrasound-guided TPVB was performed at the right T7-8, T8-9, T9-10, and T10-11 paravertebral interval under left lateral decubitus position, with 7.5 ml of medication injected into each paravertebral interval, for a total of 30 ml. Patient-controlled intravenous analgesia (PCIA) was used for postoperative analgesia, with 100mg oxycodone expended to 100ml with normal saline, 6-7ml per press with locked time of 15min and limited consumption of 12-15mg each hour based on the weight and basic situation of patient. Rescue analgesia was administered with flurbiprofenate 50 mg or tramadol 100 mg every 6 h when rest VAS score was ≥4. Cumulative consumption of 72 hours postoperatively was recorded. Quality of recovery 40 (QoR-40) score of 72 hours, pain visual analog (VAS) score from 6 hours to 3 months and sleep quality from discharge to 3 months after surgery were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* American Society of Anesthesiologist physical status I-III;
* Child-Pugh score A-B;
* Non anergic to medication used in this study;
* Optional/scheduled for liver resection;
* Approved participation before study.

Exclusion Criteria:

* Patients with contraindications for local nerve block such as spinal anatomic structure abnormality or local infection of puncture area;
* Anergic to medications used in this study;
* Patient have chronic pain;
* Patient receiving anticoagulants, opioids or have a history of narcotic abuse or alcohol abuse;
* Unable to complete postoperative pain score assessment or questionnaires or have mental disorders;
* Pregnant;
* BMI ≥30 kg/m2;
* Patient involving in other studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption of 72 hours after surgery | From discharge from post anesthesia care unit (PACU) to 72 hours postoperatively.
  Cumulative opioid consumption of 72 hours after surgery were recorded.

SECONDARY OUTCOMES:
Quality of recovery 40 (QoR-40) scores of 72 hours | From discharge from PACU to 72 hours postoperatively.
  Quality of recovery 40 (QoR-40) scores of 72 hours were recorded. In specific, QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is graded on a five-point Likert scale. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Pain visual analog (VAS) scores from 6 hours to 3 months | From 6 hours to 3 months after surgery.
  Pain visual analog (VAS) scores from 6 hours to 3 months were recorded. With a scale between 0 to 10, and the pain intensity increases as the number grows. In which 0 represent no pain and 10 represent worst pain.
Sleep quality | 3 months after surgery.
  Sleep quality up to 3 months were recorded. Pittsburgh Sleep Quality Index (PSQI) to assess sleep quality. The PSQI is a validated, self-administered questionnaire used to generate seven component scores calculated by 19 items which reflect subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime function. articipants with poor sleep quality are defined as those with a sum of the scores greater than 5 for these seven components.
Time to first opioid use | An average time is 2-3 hours after discharge from PACU.
  Time to first opioid use was recorded in each group from discharge from PACU to 72 hours after surgery.
Plasma bupivacaine concentration | From 30 minutes after local anesthetics administration to 72 hour after surgery.
  Measure plasma bupivacaine concentration after administration of local anesthetics.
Postoperative plasma inflammatory factors | From administration of local anesthesics to 72 hour after surgery.
  Measure postoperative plasma inflammatory factors (IL-6, IL-8, TNF-a) before administration of local anesthetics and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangling Wang, Ph. D, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No